CLINICAL TRIAL: NCT06854965
Title: Cohort Study on Factors Associated with the Evolution of Quality of Life Among Transgender Individuals in the French Population
Acronym: TRANSPOSE
Status: Not yet recruiting | Type: Observational
Sponsor: CNGE Conseil (Other)
Responsible Party: Sponsor
Other Study IDs: CNGE-2022-07; N°ID RCB : 2024-A00504-43 (Other: ANSM (Agence nationale de sécurité du médicament et des produits de santé))
Record Dates: First submitted 2025-02-03; First posted 2025-03-03 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Transgender Persons
Keywords: Transgender; Quality of Life (QoL)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This research focuses on identifying medical, social, and healthcare journey determinants associated with the evolution of quality of life in the transgender population at 12 months. To address the research question, it is planned to include 1,500 transgender individuals, among those attending healthcare professionals or associations in the French territory who have agreed to take on the role of investigators (professionals in healthcare or designated individuals within an association).

DETAILED DESCRIPTION:
Information Note:

1. What is the purpose of this research? This research focuses on identifying medical, social, and healthcare journey determinants associated with the evolution of quality of life in the transgender population at 12 months. To address the research question, it is planned to include 1,500 transgender individuals, among those attending healthcare professionals or associations in the French territory who have agreed to take on the role of investigators (professionals in healthcare or designated individuals within an association).
2. What does the research involve? In the proposed research, the investigators will assess quality of life through a standardized questionnaire. The investigators will analyse this quality of life in relation to various collected data concerning participants social context, medical data, mental health, transition journey, isolation and violence, as well as participants use of psychoactive substances.

   In the framework of this research, an initial questionnaire will be administered at time T0, during participants appointment (either via video call or in person) with a health mediator. A second questionnaire will be administered 6 months later during a second appointment (via video call or in person) with a health mediator. Finally, a third and final questionnaire will be administered 12 months after T0 during a final appointment (via video call or in person) with a health mediator. The aim of these various questionnaires is to assess the evolution of quality of life over a period of 12 months. Each questionnaire will take a maximum of 40 minutes to complete.
3. What is the research timeline? The expected duration of the research is 2 years, and the participation will be for 12 months. If person agree to participate in this research, the course of the research will be as follows: A health mediator will schedule a video (or if impossible, in-person) interview with participant. Health mediators are professionals whose role is dedicated to reducing social health inequalities. They create interfaces between various stakeholders in the healthcare system and individuals facing challenges in their healthcare and prevention journeys due to various vulnerabilities. The goal is to assist these individuals in engaging with and successfully navigating these pathways, while considering their living environment. The first questionnaire will then be completed: some sections will be filled out by participants, while other questions will be asked directly by the health mediator. The health mediator will contact participants subsequently to arrange the 6-month and 12-month interviews, which will proceed in the same manner.

   The maximum time between the presentation of the information note and the contact by the health mediator is 1 month.
4. What are the benefits of participation? By participating in this research, participants will contribute to a better understanding of the factors associated with the evolution of quality of life in transgender individuals. Moreover, participation in the 3 questionnaires (0, 6 months, 12 months) will entitle participant to receive a gift card worth €20 as a token of appreciation for participation.

   If there is a need to travel to complete the questionnaires in person, the travel expenses will be covered by the sponsor.
5. How will the collected data be processed for the research? As part of the research in which participants are invited to participate, processing of personal data will be carried out by CNGE Conseil, the research sponsor and data controller, to analyse the results.

This processing is necessary for conducting the research which serves the public interest mission entrusted to CNGE Conseil.

For this purpose, participants medical data and data regarding participants lifestyle habits, as well as ethnic origins or data relating to sexual life, will be transmitted to the Sponsor or to individuals or companies acting on its behalf, in France. This data will be identified by a participants data may be used for subsequent research or additional analyses related to this research in collaboration with private or public partners, in France or abroad, under conditions ensuring their confidentiality and the same level of protection as European legislation. Participants may oppose at any time to the subsequent use of participants data by contacting the qualified person who proposed participation in this research project. Participants data will be retained only for the period strictly necessary and proportionate to the purpose of the research. They will be kept in the information systems of the data controller for up to two years after the last publication of the research results.

Participants data will then be archived in accordance with applicable regulations (article R1123-63 of the French Public Health Code). The archiving of research documents will be for a minimum of 15 years.

ELIGIBILITY:
Inclusion Criteria:

* Person identifying themselves as trans
* Person of legal age (≥ 18 years)
* Person living in France
* Person who has not expressed any opposition after receiving full information about the protocol
* Person who understands and speaks French, or who is an allophone speaking English, Spanish or Portuguese

Exclusion Criteria:

* People who do not understand or speak French, English, Spanish or Portuguese.
* Person under guardianship or curatorship, under legal protection or under safeguard of justice
* Anyone who has expressed their opposition after receiving full information about the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Transgender Individuals
Study Population: Transgender Individuals
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2025-02-28 (Estimated); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Change in quality of life (WHOQOL-BREF) between 0 and 12 months. | From enrollment to the last questionnaire at 12 months
  Differences in the WHOQOL-BREF between 0 and 12 months. The WHOQOL-BREF (World Health Organization Quality Of Life tool) consists of four dimensions: physical health, psychological health, social relationships and environment, with scores ranging from 0 to 100. A higher score denotes a higher quality of life.

SECONDARY OUTCOMES:
Quality of life (WHOQOL-BREF) at baseline and 6 months | Baseline and 6 months
  WHOQOL-BREF at baseline and 6 months. The WHOQOL-BREF (World Health Organization Quality Of Life tool) consists of four dimensions: physical health, psychological health, social relationships and environment, with scores ranging from 0 to 100. A higher score denotes a higher quality of life.
Change in quality of life (WHOQOL-BREF) between 0 and 6 months. | From baseline to 6 months
  Differences in WHOQOL-BREF between 0 and 6 months. The WHOQOL-BREF (World Health Organization Quality Of Life tool) consists of four dimensions: physical health, psychological health, social relationships and environment, with scores ranging from 0 to 100. A higher score denotes a higher quality of life.
Mental health at baseline | Baseline
  Mental health assessed with MHC-SF tool
Sexual health at baseline | Baseline
  Sexual health defined by history of STIs and unprotected sexual intercourse
Addictions at baseline | Baseline
  Addictions assessed with ASSIST tool
Screenings at baseline | Baseline
  Participation in organized screenings for breast cancer, cervical cancer and colorectal cancer and individual screenings of STI
Iatrogeny at baseline | Baseline
  Complications related to hormone therapy or transition surgery
Comorbidities at baseline | Baseline
  Presence of comorbidities (cardiovascular diseases, cardiovascular risk factors, various pathologies, etc.)
Violence experienced at baseline | Baseline
  Types of violence experienced (verbal, physical, sexual, psychological, economic)
Transition modalities | At baseline, 6 months and 12 months
  Transition modalities (social transition, hormone therapy, surgery)
Healthcare pathway | At baseline, 6 months and 12 months
  Healthcare professionals consulted
Self-medication | At baseline, 6 months and 12 months
  Use of self-medication in the context of hormone therapy

CONTACTS AND LOCATIONS:
Locations (1):
- CNGE Conseil, Paris, France

IPD SHARING:
Plan to Share IPD: No